CLINICAL TRIAL: NCT03748186
Title: A Phase 1 Open-Label, Safety, Pharmacokinetic and Preliminary Efficacy Study of STRO-002, an Anti-Folate Receptor Alpha (FolRα) Antibody-Drug Conjugate (ADC), in Patients With Advanced Epithelial Ovarian Cancer (Including Fallopian Tube or Primary Peritoneal Cancers) and Endometrial Cancers
Brief Title: Study of STRO-002, an Anti-Folate Receptor Alpha (FolRα) Antibody Drug Conjugate in Ovarian & Endometrial Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sutro Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STRO-002-GM1
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma; Ovary Cancer; Endometrial Cancer; Endometrioid Adenocarcinoma; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Carcinoma, Endometrioid; Fallopian Tube Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a modified 3+3 dose escalation study with a dose expansion. Dose escalation is in advanced ovarian cancer patients with relapsed or refractory disease to standard approved therapy. Dose expansion includes 2 cancer populations, ovarian cancer and endometrial cancer. The ovarian cancer expansion cohorts are Cohort A and Cohort C. Cohort A is a dose ranging design with randomization into 2 dose levels of STRO-002, 4.3 mg/kg and 5.2mg/kg. Cohort C is a single dose cohort design, STRO-002 5.2 mg/kg with prophylactic pegfilgrastim. Dose expansion in endometrial cancer (Cohort B) is a single dose cohort design, STRO-002 5.2 mg/kg. Endometrial subjects with prior pelvic irradiation will start treatment of STRO-002 at 4.3 mg/kg with step up to 5.2 mg/kg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STRO-002 treatment (Experimental): Dose Escalation: STRO-002 at increasing dose levels
  Dose Expansion: STRO-002 at 4.3 mg/kg and 5.2 mg/kg
  Interventions: Drug: STRO-002

INTERVENTIONS:
Drug: STRO-002 — intravenous antibody drug conjugate

SUMMARY:
Phase 1 trial to study the safety, pharmacokinetics and preliminary efficacy of STRO-002 given intravenously every 3 weeks.

DETAILED DESCRIPTION:
This study is a phase 1, open-label, multicenter, dose-escalation study with dose expansion to identify the maximum tolerated dose (MTD), the recommended phase 2 dose (RP2D) and to evaluate the safety, tolerability, and preliminary antitumor activity of STRO-002 in adult subjects with advanced epithelial ovarian cancer (EOC), including fallopian or primary peritoneal cancer, and endometrial cancer. Fallopian tube and primary peritoneal cancers are treated in the same manner as epithelial ovarian cancers and are thus included in this phase 1 study. Subjects enrolled in the study will be required to have progressive or recurrent disease after standard approved therapy as defined in the study eligibility criteria. The study has completed dose escalation and is currently in dose expansion, enrolling endometrial and ovarian cancer subjects.

All subjects enrolled on the study are required to have tumor tissue for determining folate receptor alpha (FolRα) expression levels, either from a prior surgery or tumor biopsy or from a biopsy performed during study screening. The testing for FolRα is done via an ICH assay. A minimum level of FolRα expression is required for enrollment for endometrial cancer but not for ovarian cancer.

Study drug, STRO-002, is administered by intravenous (IV) infusion on day 1 of 21-day cycles. Clinical evaluations and/or laboratory tests will be performed at a pre-specified schedule-weekly for cycles 1-4, and at the beginning of every cycle starting with cycle 5 as described in the schedule of assessments. Samples for PK analysis will occur at specific times on days 1, 8, and 15 of cycles 1 and 4, Day 1 of cycles 2, 3, and 5 and at the end of treatment (EOT) visit. The study requires imaging with a CT or MRI scan of the chest abdomen and pelvis at screening, every 6 weeks after enrollment for the first 18 weeks, then every 9 weeks, and at the end of treatment (EOT) visit. Additional X-rays may be required to confirm disease responses and per local institution standard of care.

Additional clinical evaluations and lab testing may occur at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Measurable disease per RECIST 1.1
3. ECOG performance status (0-1)
4. Life expectancy > 3 months
5. Pathological confirmation of disease under study (historical information, diagnosis, pathology report, etc)

   1. Expansion Cohorts A and C: High-grade serous EOC, fallopian tube cancer or primary peritoneal cancer
   2. Expansion Cohort B: Histologically diagnosed epithelial endometrial cancer (endometrioid and serous adenocarcinomas; undifferentiated carcinoma; mixed epithelial carcinoma; or adenocarcinoma NOS)
6. Relapsed and/or progressive disease

   1. Dose Expansion Cohorts A and C (Ovarian Cancer):

      * Platinum resistant and received 1-3 prior regimens or
      * Platinum sensitive and either:
      * Progressed after 2 prior lines of platinum therapy (regardless of platinum status)and received 2-3 prior regimens or
      * Progressed after 1 line of platinum therapy and 1 line of non-platinum therapy and received a total of 2-3 prior regimens if contraindicated to receive second platinum regimen.
   2. Dose Expansion Cohort B (Endometrial Cancer):

      * Relapsed or progression after at least 1 platinum-based chemotherapy regimen or 1 immunotherapy-based regimen but not to exceed more than 3 prior regimens.
7. Fresh or archival tumor tissue samples

Exclusion Criteria:

1. Low grade (grade 1) ovarian carcinoma, clear cell, mucinous and sarcomatous ovarian carcinomas (Cohort A).
2. Endometrial carcinosarcomas, leiomyosarcoma and stromal sarcomas (Cohort B).
3. Prior treatment with a FolRα-targeting ADCs or FolRα-targeting vaccines
4. Platinum-refractory during frontline treatment (Cohorts A and C)
5. Greater than 3 lines of prior treatment
6. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy or to antibody-related fusion protein treatment
7. Preexisting clinically significant ocular disorders, clinically significant pre-exisiting ocular disorders, severe chronic obstructive pulmonary disease or asthma, clinically significant cardiac or cerebrovascular disease, or other significant concurrent, uncontrolled medical condition
8. Metastatic central nervous system or meningeal disease
9. Concurrent participation in another therapeutic treatment trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients are required to have ovarian, fallopian, primary peritoneal or endometrial cancer.
Enrollment: 136 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability of STRO-002) | 18 months
  Incidence of adverse events (AEs) observed across STRO-002 dose levels
Part 1: Define the recommended phase 2 dose (RP2D) of STRO-002 | 18 months
  Frequency of dose-limiting toxicity and exposure across STRO-002 dose levels
Part 1: Define the maximum tolerated dose (MTD) of STRO-002 | 18 months
  Frequency of dose-limiting toxicity and exposure across STRO-002 dose levels
Part 2: Evaluate preliminary anti-tumor activity (ovarian, Fallopian and primary peritoneal cancer patients) | 24 months
  Objective response rate per RECIST 1.1
Part 2: Evaluate preliminary anti-tumor activity (endometrial cancer patients) | 24 months
  Objective response rate per RECIST 1.1

SECONDARY OUTCOMES:
Part 1: Characterize the pharmacokinetics (PK) of STRO-002 by measuring the maximum plasma concentration (Cmax) | 18 months
  Measurement of maximum plasma concentration after the administration of STRO-002
Part 1: Characterize the PK of STRO-002 by measuring the half-life (t1/2) of STRO-002 | 18 months
  Measurement of terminal half-life of STRO-002 after the administration of STRO-002
Part 1: Characterize the PK of STRO-002 measuring the total area under the concentration versus time curve from zero to infinity (AUCinf) | 18 months
  Measurement of AUC to infinity (AUCinf)
Part 1: Characterize the PK of STRO-002 by measuring the clearance (CL) | 18 months
  Measurement of total body clearance
Part 1: Characterize the PK of STRO-002 by measuring the the steady state volume of distribution (Vss) | 18 months
  Measurement of steady state volume of distribution
Part 1: Assess the formulation of anti-drug antibodies to STRO-002 | 18 months
  Circulating anti-drug antibodies (ADAs) formed to STRO-002
Part 2: Further evaluate the incidence of Treatment-Emergent Adverse Events (Safety and Tolerability of STRO-002) | 24 months
  Number of patients with abnormal laboratory values and/or adverse events related to STRO-002 treatment
Part 2: Evaluate preliminary anti-tumor efficacy with a time-to-event analysis of duration of response (DOR) in patients treated with STRO-002 | 24 months
  Duration of response per RECIST 1.1
Part 2: Evaluate preliminary anti-tumor efficacy with a time-to-event analysis of progression-free survival (PFS) in patients treated with STRO-002 | 24 months
  Progression-free survival per RECIST 1.1
Part 2: Evaluate preliminary effect of STRO-002 treatment on CA-125 levels | 24 months
  Response assessment based on the Gynecologic Cancer Intergroup (GCIG) criteria
Part 2: Characterize the PK of STRO-002 by measuring the maximum plasma concentration (Cmax) | 24 months
  Measurement of maximum plasma concentration (Cmax) after the administration of STRO-002
Part 2: Characterize the PK of STRO-002 by measuring the area under the plasma concentration versus time curve (AUC) | 24 months
  Measurement of AUC to infinity (AUC inf)
Part 2: Characterize the PK of STRO-002 by measuring the clearance (CL) | 24 months
  Measurement of total body clearance

OTHER OUTCOMES:
Part 1: Preliminary assessment of the anti-tumor activity of STRO-002 | 18 months
  Objective response rate per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (27):
- United States (23):
  - Arizona Oncology - Tucson, Tucson, Arizona
  - UCLA Jonsson Comprehensive Cancer Center Clinical Research Unit, Los Angeles, California
  - Sutter Health- Palo Alto Medical Foundation, San Francisco, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Miami Cancer Institue, Baptist Health South Florida, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Augusta Oncology, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Maryland Oncology Hematology, Rockville, Maryland
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NYU Langone Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Ohio State University, James Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Cancer Care Northwest-South Spokane, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Spain (4):
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Clínica Universidad de Navarra -Madrid, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Zhou S, Abrahams CL, Krimm S, Smith J, Bajjuri K, Stephenson HT, Henningsen R, Hanson J, Heibeck TH, Calarese D, Tran C, Yin G, Stafford RL, Yam AY, Kline T, De Almeida VI, Sato AK, Lupher M, Bedard K, Hallam TJ. Discovery of STRO-002, a Novel Homogeneous ADC Targeting Folate Receptor Alpha, for the Treatment of Ovarian and Endometrial Cancers. Mol Cancer Ther. 2023 Feb 1;22(2):155-167. doi: 10.1158/1535-7163.MCT-22-0322. PMID 36459691